CLINICAL TRIAL: NCT02863926
Title: Safety and Efficacy of Concentrated Autologous Concentrated Bone Marrow Aspirate (cBMA) in Preventing Wound Complications in Below Knee Amputation (BKA) (The MarrowCHAMP Study)
Brief Title: Use of Autologous Concentrated Bone Marrow Aspirate in Preventing Wound Complications in Below Knee Amputation (BKA)
Acronym: MarrowCHAMP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Murphy (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor-Investigator, Michael Murphy, Principal Investigator, MD, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1511774456
Record Dates: First submitted 2016-05-02; First posted 2016-08-11 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Artery Disease; Vascular Disease; Critical Limb Ischemia
Keywords: BKA; amputation; MarrowStim; below knee amputation; wound complication; vascular disease; critical limb ischemia; peripheral artery disease; AKA; stem cells; bone marrow
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Autologous bone marrow derived mesenchymal stromal cells will be delivered intramuscularly in the lower extremity of participants undergoing lower extremity major amputation to assess incidence of wound healing and infection prevention.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Day 7 (Experimental): BKA performed at 7 days post autologous cBMA injection. Injection of cBMA aspirate into the index leg
  Interventions: Biological: Injection of cBMA aspirate into the index leg
- Day 14 (Experimental): BKA performed at 14 days post autologous cBMA injection. Injection of cBMA aspirate into the index leg
  Interventions: Biological: Injection of cBMA aspirate into the index leg
- Day 21 (Experimental): BKA performed at 21 days post autologous cBMA injection. Injection of cBMA aspirate into the index leg
  Interventions: Biological: Injection of cBMA aspirate into the index leg

INTERVENTIONS:
Biological: Injection of cBMA aspirate into the index leg — Injection of cBMA into the anterior tibialis muscle and upper index leg of subjects scheduled for semi-elective BKA 7-21 days before surgery
  Other Names: concentrated bone marrow; cBMA

SUMMARY:
Patients scheduled for major extremity lower amputation to receive bone marrow cells (cBMA) injected IM in the leg proximal to the amputation in the index limb to prevent ischemic wound complications after surgery.

DETAILED DESCRIPTION:
Patients scheduled for amputation will receive bone marrow cells concentrated via the MarrowStim device (cBMA) injected IM at 25 sites in the leg proximal to the amputation in the index limb to prevent ischemic wound complications after surgery. cBMA will be injected into the anterior tibialis muscle below the point of amputation in an area approximately 3cm^2 x 2cm^2 for analytical purposes. Patients will be scheduled for amputation at Days 7, 14, or 21 post injection. Safety will be evaluated by review of treatment related adverse events (AE) during the 52-week follow-up period. The investigator will compare rates of wound complications and amputation revisions to historical controls at the institution to assess trends in therapeutic efficacy.

Patients will undergo amputation and injection sites will be harvested at that time. Immunohistochemical staining (IHC) will determine capillary density and local host immune responses. Angiogenic and inflammatory cytokines will be quantified using a multiplex array system and quantitative polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 40 and ≤90 years of age.
2. Patients requiring below knee amputation, as determined by an independent vascular specialist.
3. If ulceration or gangrene present, it is distal to malleoli (to allow adequate length of ATM for 4 injections 4 cm. apart)
4. BKA can safely be performed up to 30 days after screening, as determined by an independent vascular or orthopedic surgeon. This information will be documented in subjects' case report forms (CRFs).
5. Females of childbearing potential must be willing to use one form of birth control for the duration of the study. Female participants must undergo a blood or urine pregnancy test at screening.

Exclusion Criteria:

1. Patients who are pregnant, planning to become pregnant in the next 12 months, or lactating.
2. Significant hepatic dysfunction (ALT or AST greater than 2 times normal).
3. CHF hospitalization within the last 1 month prior to enrollment.*
4. Acute coronary syndrome (ACS) in the last 1 month prior to enrollment.*
5. HIV positive, or active, untreated HCV.
6. History of cancer within the last 5 years, except basal cell skin carcinoma
7. Any bleeding diathesis defined as an INR ≥ 2.0 (off anticoagulation therapy) or history of platelet count less than 70,000 or hemophilia.
8. Inability to provide written informed consent due to cognitive or language barriers (interpreter permitted).
9. Concurrent enrollment in another clinical investigative trial.
10. Any condition requiring immunosuppressant medications (e.g., for treatment of organ transplants, psoriasis, Crohn's disease, alopecia areata).
11. Presence of any clinical condition that in the opinion of the PI or the sponsor makes the patient not suitable to participate in the trial.

    * As defined by the standard definitions of CHF and ACS by the American Heart Association.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Murphy, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with investigators at the Indiana University School of Medicine as well as at other collaborating institutions.
Supporting Information: CSR
Time Frame: Data will become available as it is generated and will be available for future, yet-to-be-written protocols.
Access Criteria: Access to de-identified data will be granted for future PI approved indications.

REFERENCES:
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Santilli JD, Santilli SM. Chronic critical limb ischemia: diagnosis, treatment and prognosis. Am Fam Physician. 1999 Apr 1;59(7):1899-908. PMID 10208708
- [Background] Albers M, Fratezi AC, De Luccia N. Assessment of quality of life of patients with severe ischemia as a result of infrainguinal arterial occlusive disease. J Vasc Surg. 1992 Jul;16(1):54-9. PMID 1619725
- [Background] Huang PP, Li SZ, Han MZ, Xiao ZJ, Yang RC, Qiu LG, Han ZC. Autologous transplantation of peripheral blood stem cells as an effective therapeutic approach for severe arteriosclerosis obliterans of lower extremities. Thromb Haemost. 2004 Mar;91(3):606-9. doi: 10.1160/TH03-06-0343. PMID 14983238
- [Background] Cruz CP, Eidt JF, Capps C, Kirtley L, Moursi MM. Major lower extremity amputations at a Veterans Affairs hospital. Am J Surg. 2003 Nov;186(5):449-54. doi: 10.1016/j.amjsurg.2003.07.027. PMID 14599605
- [Background] Dillingham TR, Pezzin LE, MacKenzie EJ. Limb amputation and limb deficiency: epidemiology and recent trends in the United States. South Med J. 2002 Aug;95(8):875-83. doi: 10.1097/00007611-200208000-00018. PMID 12190225
- [Background] Dillingham TR, Pezzin LE, Shore AD. Reamputation, mortality, and health care costs among persons with dysvascular lower-limb amputations. Arch Phys Med Rehabil. 2005 Mar;86(3):480-6. doi: 10.1016/j.apmr.2004.06.072. PMID 15759232
- [Background] Castronuovo JJ Jr, Deane LM, Deterling RA Jr, O'Donnell TF Jr, O'Toole DM, Callow AD. Below-knee amputation: is the effort to preserve the knee joint justified? Arch Surg. 1980 Oct;115(10):1184-7. doi: 10.1001/archsurg.1980.01380100032007. PMID 7425829
- [Background] Nehler MR, Coll JR, Hiatt WR, Regensteiner JG, Schnickel GT, Klenke WA, Strecker PK, Anderson MW, Jones DN, Whitehill TA, Moskowitz S, Krupski WC. Functional outcome in a contemporary series of major lower extremity amputations. J Vasc Surg. 2003 Jul;38(1):7-14. doi: 10.1016/s0741-5214(03)00092-2. PMID 12844082
- [Background] Lim TS, Finlayson A, Thorpe JM, Sieunarine K, Mwipatayi BP, Brady A, Abbas M, Angel D. Outcomes of a contemporary amputation series. ANZ J Surg. 2006 May;76(5):300-5. doi: 10.1111/j.1445-2197.2006.03715.x. PMID 16768686
- [Background] Prockop DJ. Repair of tissues by adult stem/progenitor cells (MSCs): controversies, myths, and changing paradigms. Mol Ther. 2009 Jun;17(6):939-46. doi: 10.1038/mt.2009.62. Epub 2009 Mar 31. PMID 19337235
- [Background] Markel TA, Wang Y, Herrmann JL, Crisostomo PR, Wang M, Novotny NM, Herring CM, Tan J, Lahm T, Meldrum DR. VEGF is critical for stem cell-mediated cardioprotection and a crucial paracrine factor for defining the age threshold in adult and neonatal stem cell function. Am J Physiol Heart Circ Physiol. 2008 Dec;295(6):H2308-14. doi: 10.1152/ajpheart.00565.2008. Epub 2008 Oct 10. PMID 18849336
- [Background] Kinnaird T, Stabile E, Burnett MS, Shou M, Lee CW, Barr S, Fuchs S, Epstein SE. Local delivery of marrow-derived stromal cells augments collateral perfusion through paracrine mechanisms. Circulation. 2004 Mar 30;109(12):1543-9. doi: 10.1161/01.CIR.0000124062.31102.57. Epub 2004 Mar 15. PMID 15023891
- [Background] Seok J, Warren HS, Cuenca AG, Mindrinos MN, Baker HV, Xu W, Richards DR, McDonald-Smith GP, Gao H, Hennessy L, Finnerty CC, Lopez CM, Honari S, Moore EE, Minei JP, Cuschieri J, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Jeschke MG, Klein MB, Gamelli RL, Gibran NS, Brownstein BH, Miller-Graziano C, Calvano SE, Mason PH, Cobb JP, Rahme LG, Lowry SF, Maier RV, Moldawer LL, Herndon DN, Davis RW, Xiao W, Tompkins RG; Inflammation and Host Response to Injury, Large Scale Collaborative Research Program. Genomic responses in mouse models poorly mimic human inflammatory diseases. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3507-12. doi: 10.1073/pnas.1222878110. Epub 2013 Feb 11. PMID 23401516
- [Background] Deutsch MA, Sturzu A, Wu SM. At a crossroad: cell therapy for cardiac repair. Circ Res. 2013 Mar 15;112(6):884-90. doi: 10.1161/CIRCRESAHA.112.275974. No abstract available. PMID 23493304
- [Background] Wang L, Cao L, Shansky J, Wang Z, Mooney D, Vandenburgh H. Minimally invasive approach to the repair of injured skeletal muscle with a shape-memory scaffold. Mol Ther. 2014 Aug;22(8):1441-1449. doi: 10.1038/mt.2014.78. Epub 2014 Apr 28. PMID 24769909
- [Background] Murphy MP, Lawson JH, Rapp BM, Dalsing MC, Klein J, Wilson MG, Hutchins GD, March KL. Autologous bone marrow mononuclear cell therapy is safe and promotes amputation-free survival in patients with critical limb ischemia. J Vasc Surg. 2011 Jun;53(6):1565-74.e1. doi: 10.1016/j.jvs.2011.01.074. Epub 2011 Apr 22. PMID 21514773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were invited to participate in the study on a first-come basis, recruited from the Investigator's patient population and by referrals from other physicians who have patients recommended for major amputation. The study team received referrals after the patient was seen by their own vascular or orthopedic specialist and the amputation was recommended to them.
Pre-assignment Details: Of 7 screened patients, 6 met inclusion criteria and were treated.
Period: Overall Study
Arm/Group | Day 7 | Day 21
Started | 5 | 1
Per Protocol Population Week 6 | 4 | 1
Per Protocol Population Week 52 | 3 | 0
Completed | 3 | 0
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: One patient randomized into the Day 7 arm/group could not tolerate their leg pain and had amputation 3 days after BMAC treatment.
  No participants had an interval of 14 days from BMAC injection to below knee amputation date.
Groups:
- Total: Total of all reporting groups
Arm/Group | Day 7 | Day 21 | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (5.57) | 66 (0) | 63 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Current Smoker [Number; unit: participants] | 4 | 1 | 5
Diabetes Mellitus [Number; unit: participants] | 5 | 1 | 6
Hgb A1C % [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 9.04 (1.46) | 8.0 (0) | 8.52 (0.52)
Systolic Blood Pressure [Mean (Standard Deviation); unit: Pressure during heartbeat in mmHg] | 122 (27.6) | 187 (0) | 133 (35.0)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: Pressure between heartbeats in mmHg] | 68.8 (71.5) | 85 (0) | 71.5 (9.2)
Body Mass index (BMI) [Mean (Standard Deviation); unit: weight in kg/height in meters^2] | 31.62 (3.41) | 24.5 (0) | 30.43 (4.09)
eGFR [Mean (Standard Deviation); unit: Renal filtration rate in mg/mmol] | 61.96 (36.1) | 52 (0) | 60.3 (33.17)
Index Leg TcPO2 [Mean (Standard Deviation); unit: Oxygen level at skin in mmHg] | 35.25 (21.69) | 0 (0) | 35.25 (21.69)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events Occurring During the Enrollment Period as Assessed by the Investigator Using the CTCAE 4.0 Scale.
Description: Safety will be evaluated by review of treatment related AEs during the 12-month follow-up period. The study will be terminated in the event of a Grade 4-5 unexpected event based on the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Treatment-related AEs will be categorized overlapping systems and severities. Three categories of systems are cardiovascular, respiratory, or infectious. Two categories of severity will be serious adverse (SAE) and major adverse cardiac events (MACE). Binomial confidence Intervals at the 95% confidence level and p-values for these 3 groups will be calculated. Since previous trials have not reported AEs with cBMA treatment, confidence intervals will be generated by the method of the Wilson Score Interval.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Day 7 | Day 21
Number analyzed (Participants) | 5 | 1
Participants | 2 | 0

2. Secondary Outcome: Number of Participants With Conversion From Below Knee Amputation to Above Knee Amputation as Evidenced by Wound Complications at the Below Knee Amputation Stump Site.
Description: Documentation will be collected on wound complications at the below knee amputation surgical site resulting in necessity of revision/conversion to above knee amputation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Day 7 | Day 21
Number analyzed (Participants) | 5 | 1
Participants | 0 | 0

3. Secondary Outcome: The Role of Autologous Bone Marrow Cells Injected in Human Skeletal Muscle in Inducing Capillary Vessel Formation at the Time of Below Knee Amputation.
Description: Continuous confidence intervals at the 95% level will be constructed to explore differences among the time-tiered administration of MSC for the quantity of capillary density in muscle fibers.
Time Frame: 12 months
Population: Immunostaining for the CD31 antigen was selected to measure the capillary density, reported as CD31-positive features normalized to fiber number. For capillary density quantification, CD31 positive profiles were counted using a custom algorithm and nuclei were counted using a pipeline that we designed in CellProfiler.
Measure: Mean (Standard Error); unit: CD31-positive capillaries/fiber
Arm/Group | Day 7 | Day 21
Number analyzed (Participants) | 5 | 1
CD31-positive capillaries/fiber
  Proximal ATM Segment A | 1.089 (0.052) | 1.431 (0.553)
  Distal ATM Segment B | 1.373 (0.050) | 1.673 (0.232)
  Distal ATM Segment C | 1.064 (0.056) | 1.526 (0.508)
  Distal ATM Segment D | 1.065 (0.064) | 1.197 (0.460)
  Control Segment - Soleus | 1.191 (0.104) | NA (NA) — For this one patient in "Day 21" group, we did not have enough appropriate soleus tissue specimen for completing the ICC analysis.

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Day 7 | Day 21
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/5 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 7 (N=5) | Day 21 (N=1)
Wound dehiscence at amputation site (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Fascial disruption or dehiscence without evisceration; primary wound closure or revision by operative intervention indicated
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2) | 0 (0) — Diabetic ketoacidosis
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral ischemia, non-index leg (Vascular disorders) | 1 (1) | 0 (0) — Recurrent or prolonged ischemia in the non-treated lower extremity
Wound infection, non-index leg (Infections and infestations) | 1 (1) | 0 (0) — Presence of wound/ulcer in the non-treated lower extremity
Major amputation, non-index leg (Vascular disorders) | 1 (1) | 0 (0) — Amputation below the knee of non-treated lower extremity
Depression, worsening (Psychiatric disorders) | 0 (0) | 1 (1)
Seroma at amputation site, index leg (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Seroma formation at surgical site after below knee amputation
Chronic kidney disease with acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) — CKD Stage III
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Above Knee Amputation (Vascular disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 7 (N=5) | Day 21 (N=1)
Pain at amputation site (General disorders) | 4 (4) | 0 (0) — Pain experienced at the surgical amputation site
Wound developed on non-index foot (Vascular disorders) | 1 (1) | 0 (0) — Wounds, ulcers occurring on the non-treated lower extremity
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Oral Candidiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic anemia, worsening (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Wound, non-index extremity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Wound development to non-treated lower extremity
Chronic hypertension, worsening (Cardiac disorders) | 0 (0) | 1 (1)
Fever of unknown origin (General disorders) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 0 (0) | 1 (2)
Skin integrity worsening, amputation site (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Iliac crest pain, post bone marrow aspiration (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
COVID-19 research activities Hold leading to slower enrollment and Cost-prohibitive to resume enrollment at VA for additional participants leading to early closure of study and low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02863926/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02863926/ICF_001.pdf